CLINICAL TRIAL: NCT00450502
Title: A Phase I Study of Batracylin (NSC320846) in Subjects With Solid Tumors and Lymphomas
Brief Title: Safety of Batracylin in Patients With Solid Tumors and Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 070097; 07-C-0097; NCT01445184 (obsolete NCT alias)
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2013-08-14

CONDITIONS: Neoplasms
Keywords: Cytotoxic; Pharmacokinetics; Toxicity; Neoplasms; Pharmacogenomics; Solid Tumor; Lymphoma
MeSH Terms: conditions — Neoplasms; Lymphoma | interventions — batracylin

INTERVENTIONS:
Drug: Batracylin

SUMMARY:
Background:

* Batracylin advanced through the National Cancer Institute (NCI) drug development pipeline until its evaluation at Stage 3 on July 1989, It was then proposed for a phase I investigation based on its activity against as TOPO II inhibitor in s.c. mouse colon 38, PANC03, COLO9, and cisplatin- and doxorubicin-resistant P388 tumors.
* IND-directed oral toxicology studies indicated interspecies variation in toxicity. Rats were found to be highly sensitive to batracylin. Ames et al showed that the interspecies variation in toxicity was consistent with the pattern of metabolism of the compound by N-acetyltransferase 2 (NAT2) to the acetylated form, N-Ac-batracylin, (a highly toxic molecule)
* We hypothesize that batracylin can be administered safely in slow acetylator NAT2 genotype patients and can be rapidly evaluated for its potential as a tumor-suppressing agent.

Objectives:

* Define the maximum tolerated dose, dose-limiting toxicities, and toxicity profile associated with the oral administration of batracylin daily x7 consecutive days, repeated every 28 days in patients with solid tumors and lymphomas.
* Define the pharmacokinetics of oral batracylin administered daily x7 consecutive days every 28 days.
* Obtain preliminary evidence of anti-tumor activity of batracylin in patients with solid tumors or lymphoma.
* Correlate polymorphisms in slow acetylators NAT2 genotypes (NAT2 5, NAT2 6, NAT2 7, and NAT2 14) with pharmacokinetics results.
* Evaluate the inter-subject variability and toxicity ratio, (N-Ac-Batra) / (batracylin).
* Evaluate the effect of batracylin treatment on gamma-H2AX levels in tumor biopsies.

Eligibility:

* Patients must have a slow acetylator NAT2 genotype defined as NAT2 5, NAT2 6, NAT2 7, or NAT2 14.
* Patients with advanced, histologically confirmed malignancies refractory to standard therapy, or those for whom no standard therapy exists.
* Patients should have adequate liver, renal, and bone marrow function.

Study Design:

* In accordance with the accelerated titration design 4B[3], dose levels will initially be increased at 100% increments, and one new patient per dose level will be treated according to a 4-week course.
* The accelerated phase ends when one patient experiences dose limiting toxicity (DLT) during the first course of treatment, or when two different patients experience grade 2, batracylin-related toxicity during the first course of treatment, or when the N-acetyl-batra AUC value reach 0.33 uM-Hour (i.e., the lower end of the range in the rat).
* When the first instance of grade 2 batracylin-related toxicity is observed, two additional patients must have been treated at that dose, or a higher dose (during any course), without experiencing moderate (grade 2) or worse (grade 3) toxicity, in order for the accelerated phase to continue.
* When the accelerated phase ends, the dose-escalation will revert to a more conservative, modified Fibonacci scheme with 40% dose-step increments, with at least 3 patients treated per dose level.

DETAILED DESCRIPTION:
Background:

* Batracylin advanced through the National Cancer Institute (NCI) drug development pipeline until its evaluation at Stage 3 on July 1989, It was then proposed for a phase I investigation based on its activity against as TOPO II inhibitor in s.c. mouse colon 38, PANC03, COLO9, and cisplatin- and doxorubicin-resistant P388 tumors.
* IND-directed oral toxicology studies indicated interspecies variation in toxicity. Rats were found to be highly sensitive to batracylin. Ames et al showed that the interspecies variation in toxicity was consistent with the pattern of metabolism of the compound by N-acetyltransferase 2 (NAT2) to the acetylated form, N-Ac-batracylin, (a highly toxic molecule)
* We hypothesize that batracylin can be administered safely in slow acetylator NAT2 genotype patients and can be rapidly evaluated for its potential as a tumor-suppressing agent.

Objectives:

* Define the maximum tolerated dose, dose-limiting toxicities, and toxicity profile associated with the oral administration of batracylin daily for 7 consecutive days, repeated every 28 days in patients with solid tumors and lymphomas.
* Define the pharmacokinetics of oral batracylin administered daily for 7 consecutive days every 28 days.
* Obtain preliminary evidence of anti-tumor activity of batracylin in patients with solid tumors or lymphoma.
* Correlate polymorphisms in slow acetylators NAT2 genotypes (NAT2 5, NAT2 6, NAT2 7, and NAT2 14) with pharmacokinetics results.
* Evaluate the inter-subject variability and toxicity ratio, (N-Ac-Batra) / (batracylin).
* Evaluate the effect of batracylin treatment on gamma-H2AX levels in tumor biopsies.

Eligibility:

* Patients must have a slow acetylator NAT2 genotype defined as NAT2 5, NAT2 6, NAT2 7, or NAT2 14.
* Patients with advanced, histologically confirmed malignancies refractory to standard therapy, or those for whom no standard therapy exists.
* Patients should have adequate liver, renal, and bone marrow function.

Study Design:

* In accordance with the accelerated titration design 4B[3], dose levels will initially be increased at 100% increments, and one new patient per dose level will be treated according to a 4-week course.
* The accelerated phase ends when one patient experiences dose limiting toxicity (DLT) during the first course of treatment, or when two different patients experience grade 2, batracylin-related toxicity during the first course of treatment, or when the N-acetyl-batra AUC value reach 0.33 uM-Hour (i.e., the lower end of the range in the rat).
* When the first instance of grade 2 batracylin-related toxicity is observed, two additional patients must have been treated at that dose, or a higher dose (during any course), without experiencing moderate (grade 2) or worse (grade 3) toxicity, in order for the accelerated phase to continue.
* When the accelerated phase ends, the dose-escalation will revert to a more conservative, modified Fibonacci scheme with 40% dose-step increments, with at least 3 patients treated per dose level.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Patients must have histologically confirmed (by the NIH pathology department) solid tumor malignancy or lymphoma that is metastatic or unresectable for which standard curative measures do not exist, or are associated with minimal patient survival benefit.
2. Patients must have measurable or evaluable disease.
3. Patients must have completed any chemotherapy or biologic therapy greater than or equal to 4 weeks prior to entering the study (6 weeks for nitrosoureas or mitomycin C, or UCN-01). Patients must be greater than or equal to 2 weeks since any prior administration of study drug in a exploratory IND/Phase Zero study. Patients must be greater than or equal to 1 month since any prior radiation or major surgery. Patients must have recovered to eligibility levels from prior toxicity or adverse events. However, patients receiving bisphosphonates for any cancer or undergoing androgen deprivation therapy for prostate cancer are eligible for this therapy.
4. Age greater than or equal to 18 years.
5. The Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2 (Karnofsky greater than or equal to 60%).
6. Life expectancy greater than 3 months.
7. Patients must have normal or adequate organ and marrow function as defined below:

   * Absolute neutrophil count greater than or equal to 1,500/microL.
   * Platelets greater than or equal to 100,000/microL.
   * Total bilirubin within less than or equal to 1.5 normal institutional limits.
   * AST (SGOT)/ALT (SGPT) less than or equal to 2.5 x institutional upper limit of normal.
   * creatinine less than 1.5 x upper limit of normal

   OR

   -creatinine clearance greater than or equal to 60 mL/min/1.73 m(2) for patients with creatinine levels greater than or equal to 1.5 times upper limit of normal.

   We will allow patients with Gilbert s syndrome with total bilirubin up to 2.5 mg/dL.
8. The effects of batracylin on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry, for the duration of study participation, and for 2 months after discontinuation from the study. Women of child bearing potential must have a negative pregnancy test in order to be eligible. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with batracylin, breastfeeding should be discontinued if the mother is treated with batracylin.
9. Patients must have a slow acetylator NAT2 genotype defined as NAT2 5, NAT2 6, NAT2 7, or NAT2 14. Theoretically slow acetylators will have lower Ac-BAT concentrations. A number of different polymorphisms in the NAT2 give rise to amino acid substitutions, and these have been demonstrated to result in absence of catalytic activity in vitro (http://www.louisville.edu/medschool/pharmacology/NAT.html). Screening for the four variant alleles (NAT2 5, NAT2 6, NAT2 7 and NAT2 14) results in the detection of the vast majority of Caucasian slow acetylators, though additional alleles are also common in other ethnic groups. The precise percentage of slow acetylators also varies with ethnic origin, ranging from 90% in North Africans to less than 10% in many Asian populations, with a frequency of 50% in Caucasians. The incidence of fast acetylators (potentially with increased toxicity) is as follow: 50% among Caucasians, 50% among Africans, 90% among Japanese, and 20% among Egyptians. We plan to select the slow acetylators NAT2 subjects and determine the batracylin MTD in this population. The screening will occur prior to the study start and before patients sign the informed consent form. Cogenics will be performing the NAT2 analysis.
10. Ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

1. Patients receiving any other investigational agents.
2. Patients with known brain metastases are excluded from this clinical trial, with the exception of patients whose brain metastatic disease status has remained stable for greater than or equal to 6 months after treatment of the brain metastases, without steroids or anti-seizure medications. These patients may be enrolled at the discretion of the principal investigator.
3. Patients with clinically significant illnesses which could compromise participation in the study, including, but not limited to, active or uncontrolled infection, immune deficiencies or confirmed diagnosis of HIV infection, Hepatitis B, Hepatitis C, uncontrolled diabetes, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Inclusion of Women and Minorities

Both men and women, and members of all races and ethnic groups, are eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-02-24; Primary Completion 2011-04-24 (Actual); Study Completion 2011-04-24 (Actual)

PRIMARY OUTCOMES:
Define the maximum tolerated dose of batracylin administered daily x7 consecutive days, repeated every 28 days in slow acetylator NAT2 genotype (NAT2 5, NAT2 6, NAT2 7, or NAT2 14) patients with solid tumors and lymphomas.

SECONDARY OUTCOMES:
Obtain preliminary evidence of anti-tumor activity of batracylin in patients with solid tumors or lymphoma.

CONTACTS AND LOCATIONS:
Overall Officials: Shivaani Kummar, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ames MM, Mathiesen DA, Reid JM. Differences in N-acetylation of the experimental antitumor agent batracylin in the mouse and the rat. Invest New Drugs. 1991 Aug;9(3):219-25. doi: 10.1007/BF00176974. PMID 1783521
- [Background] Stevens GJ, Burkey JL, McQueen CA. Toxicity of the heterocyclic amine batracylin: investigation of rodent N-acetyltransferase activity and potential contribution of cytochrome P450 3A. Cell Biol Toxicol. 2000;16(1):31-9. doi: 10.1023/a:1007692503817. PMID 10890504
- [Background] Simon R, Freidlin B, Rubinstein L, Arbuck SG, Collins J, Christian MC. Accelerated titration designs for phase I clinical trials in oncology. J Natl Cancer Inst. 1997 Aug 6;89(15):1138-47. doi: 10.1093/jnci/89.15.1138. PMID 9262252